CLINICAL TRIAL: NCT02884167
Title: Multidimensional Risk Factor Assessment in Constipation
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: ReDA-010666 QM
Record Dates: First submitted 2016-06-29; First posted 2016-08-30 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2016-08

CONDITIONS: Constipation; Risk Factors
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Patients with constipation
- Healthy individuals without constipation

SUMMARY:
Constipation is a symptom based disorder with a prevalence of 15% in the adult population and its management remains challenging. Although not life threatening, constipation is associated with impaired quality of life, increased healthcare costs and excess work absenteeism. Constipation represents a heterogeneous disorder with a multifactorial pathogenesis. Several risk factors have been suggested to lead to the condition and are divided in 3 main categories: a) physiological, b) environmental and c) demographic. To date, there is lack of large epidemiological studies on proposed aetiological factors of constipation, especially studies assessing all proposed risk factors of constipation together.

The overall aim of this study is to investigate the multidimensional (physiological, environmental and demographic) predictors of constipation with the use of a multivariate analysis statistical model.

This is a large single centre case control study comparing constipated adults with healthy individuals matched for age, gender and ethnicity.

The duration of the study is 2 weeks in total and includes a screening visit, a 2 week run-in period and a baseline visit at the end of the run-in period. Transit time between constipated and healthy individuals is assessed at baseline visit. Differences in gastrointestinal symptoms, dietary intake as well as differences in stool output (e.g. stool frequency and consistency) between constipated and healthy individuals are assessed over the baseline period (the week before the baseline visit). Differences in female sex hormone levels as well as stool markers and markers of fermentation (e.g. fecal water, stool pH, short chain fatty acids) between constipated and healthy individuals are assessed at baseline visit. Furthermore, differences in environmental measures (physical activity, anxiety, smoking) and differences in demographic measures (age, gender, body mass index) between patients suffering from constipation and healthy individuals are also assessed at baseline visit.

ELIGIBILITY:
Inclusion criteria for cases:

* Adult men or women (18-65 years)
* Symptoms of constipation for a minimum of 3 months
* Recruitment based on simplified core ROME III diagnostic criteria for functional constipation
* Average Bristol stool type of 1-4 AND frequency of 1-3 spontaneous bowel movements per week
* Cleveland Clinic constipation score (CCCS) of 8-15

Inclusion criteria for controls:

* Adult men or women (18-65 years)
* Healthy individuals without any coexisting acute or chronic disease
* Not meeting simplified core ROME III diagnostic criteria for functional constipation
* Average Bristol stool type of 2-5 AND frequency of 3-21 spontaneous bowel movements per week
* Cleveland Clinic constipation score (CCCS) of < 8

Exclusion criteria for both cases and controls:

* Pregnant or breastfeeding women
* Ongoing other diagnosed gastrointestinal disease or complication
* Alarm features such as sudden weight loss, rectal bleeding, recent change in bowel habit (<3 months), abdominal pain and stool positive for occult blood
* Prior GI surgery except cholecystectomy, appendicectomy and simple vaginal hysterectomy
* Neurologic diseases
* Ongoing therapy with drugs known to affect gut motility
* Subjects with comorbid illnesses such as cardiovascular, endocrine, renal or other chronic disease likely to affect gut motility or limit normal functions
* Self-reported symptoms of pelvic organ prolapse
* Moderate or severe active local anorectal problems
* Incapacity to consent
* Aged under 18 or over 65 years
* Any inclusion criteria listed above not met

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 patients with constipation (cases) and 100 healthy individuals without constipation (controls)
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Whole gut transit time | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary University of London, London, United Kingdom